CLINICAL TRIAL: NCT04241081
Title: Interrupting Prolonged Sitting With Periodic Interval Exercise: Effect on Postprandial Lipemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2019-10-0091
Record Dates: First submitted 2020-01-21; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Sedentary Behavior; Hypertriglyceridemia
MeSH Terms: conditions — Sedentary Behavior; Hypertriglyceridemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group-no exercise (No Intervention): A no-exercise control. Must maintain <4,500 steps per day for 3 consecutive days followed by a high fat tolerance test on day 4.
- Exercise intervention 1 (Experimental): Two consecutive days of <4,500 steps per day followed by an intervention day on day 3. Intervention day consists of interrupting 8-hour sit with bike sprint protocol every 2 hours. Participants must aim to maintain <2,500 steps on intervention day. A high fat tolerance test will be performed the following day on day 4.
  Interventions: Behavioral: Interrupting Prolonged Sitting with Periodic Interval Exercise: Effect on Postprandial Lipemia
- Exercise intervention 2 (Experimental): Two consecutive days of <4,500 steps per day followed by an intervention day. Intervention day consists of interrupting 8-hour sit with bike sprint protocol every 6 hours. Participants must aim to maintain <2,500 steps on intervention day. A high fat tolerance test will be performed the following day on day 4.
  Interventions: Behavioral: Interrupting Prolonged Sitting with Periodic Interval Exercise: Effect on Postprandial Lipemia

INTERVENTIONS:
Behavioral: Interrupting Prolonged Sitting with Periodic Interval Exercise: Effect on Postprandial Lipemia — This is a behavioral intervention designed to determine the effect of breaking up prolonged bouts of sitting every 2 hours and every 6 hours with 5 sets of 4 second bouts of maximum effort bicycle ergometer accelerations compared to sitting alone on the blood triglyceride response and whole body fat oxidation after a high fat meal.
  Arms: Exercise intervention 1; Exercise intervention 2

SUMMARY:
Investigating the effects of interrupting various lengths of prolonged sitting with bike sprints on post prandial lipemia the next day. We will conduct three trials, one control, one with two-hour sitting intervals (total of 4 bouts of bike sprints) and one with 6-hour sitting intervals I total of two bouts of bike sprints). A milkshake high fat tolerance test will be conducted the next day and whole body fat oxidation as well as triglyceride area under the curve will be measured every hour for the duration of the 6-hour test.

ELIGIBILITY:
Inclusion Criteria:

* Inactive or recreational healthy adults aged 18-65 years old.

Exclusion Criteria:

* Lactose intolerance, cardiovascular or metabolic diagnoses, medications for cardiovascular or metabolic diagnoses, orthopedic issues barring cycling.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Triglyceride area under the curve | 6 hour long high fat tolerance test
  Blood measurements baseline and every hour during a high fat tolerance test.

SECONDARY OUTCOMES:
Whole body fat oxidation | 10 min, baseline, 2 hours post ingestion of shake, 4 hours, 6 hours.
  Expired gas collection and measurement of expired gas concentrations in mass spectrometer, baseline and every two hours during high fat tolerance test.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas, Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided